CLINICAL TRIAL: NCT01127295
Title: Breast Cancer Adjuvant Hormonotherapy : Tamoxifen and the Anti-aromatases Pharmacokinetics, Correlation With the Pharmacogenetic Characteristics PHACS Protocol : Pharmacology of Adjuvant Hormonotherapy in Breast Cancer
Brief Title: Pharmacology of Adjuvant Hormonotherapy in Breast Cancer
Acronym: PHACS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Institut Claudius Regaud (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09 SEIN 09
Record Dates: First submitted 2010-05-18; First posted 2010-05-20 (Estimated); Last update posted 2018-03-02 (Actual); Status verified 2018-03

CONDITIONS: Hormono-depending Adjuvant Breast Cancer
Keywords: Pharmacokinetics; Pharmacogenetic; tamoxifen; anti-aromatases; breast cancer; pharmacodynamy; Observance
MeSH Terms: conditions — Breast Neoplasms | interventions — Tamoxifen; Letrozole; Anastrozole; exemestane

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Tamoxifen, Anastrozole, letrozole, Exemestane (Other): Current hormonotherapy treatment in hormono dependent breast cancer
  Interventions: Drug: Tamoxifen, Letrozole, Anastrozole or Exemestane

INTERVENTIONS:
Drug: Tamoxifen, Letrozole, Anastrozole or Exemestane — Tamoxifen 20 mg/day during 5 years Létrozole 2.5 mg/day during 5 years Anastrozole 1 mg/day during 5 years Exémestane 25 mg/day during 5 years

SUMMARY:
This is a biomedical study of interventional type, multicenter, inter-regional.

Patients with hormono-depending breast cancer, for which an indication of adjuvant hormonotherapy treatment (according to the current treatments) was retained, will be enrolled in this study. The main objective is to estimate the correlations between pharmacokinetic and pharmacogenetic parameters of adjuvant hormonal breast cancer treatment, during the first 3 years.

ELIGIBILITY:
Inclusion Criteria:

1. Patient of more than 18 years old (menopaused or not)
2. Invasive breast cancer non-metastatic locally controlled by surgery with or without radiotherapy. Previous treatment with chemotherapy is allowed including trastuzumab
3. Cancer hormone-expressing ER and / or PR (> 10% tumor cells in Technical HIC)
4. Having a staging exploring bone, liver, lung and showing no abnormality secondary (for sub-centimeter tumors, the staging is not necessary)
5. WHO <2
6. Before the initiation of adjuvant hormonal therapy (tamoxifen, anastrozole, letrozole or exemestane) and whatever the approach chosen by the investigator (5 years of tamoxifen, 5 years of anti-aromatase or sequential patterns)
7. signed Consent collected before any specific procedure in the study
8. Patient member in a national insurance scheme.

Exclusion Criteria:

1. Patient previously treated for breast cancer receiving hormonal therapy with tamoxifen, anastrozole, letrozole or exemestane regardless of the scheme
2. Metastatic Breast cancer
3. History of another cancer diagnosed within 5 years before or uncontrolled except carcinoma in situ of cervix carcinoma, nonmelanoma skin, breast cancer (in this case, treatment with hormone therapy should be stopped for at least 6 months)
4. Any other medical or psychiatric condition or laboratory abnormality severe acute or chronic making the inclusion of the patient in the study inappropriate in the opinion of the investigator
5. Patient unable to follow procedures, visits, examinations described in the study
6. Pregnant women or nursing mothers can not participate in the study
7. Women of childbearing age must use effective contraception at study entry and up to at least three months after the end of treatment
8. Patient under legal guardianship

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Actual)
Dates: Start 2010-06-17 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2017-12-01 (Actual)

PRIMARY OUTCOMES:
Correlation between pharmacokinetic and pharmacogenetic parameters | 9 years
  To estimate the correlations between pharmacokinetic and pharmacogenetic parameters of hormonal adjuvant breast cancer treatment during the first 3 years.

SECONDARY OUTCOMES:
To estimate the relation between plasmatic concentrations, pharmacogenetic characteristic and adverse effects. | 9 years
To estimate the relation between the genetic polymorphisms and premature relapses in the first 3 years of treatment | 9 years
To estimate the link between plasmatic concentrations and the premature relapse (in the first 3 years) | 9 years
To estimate the declared therapeutic observance to the real exposure at the treatment measured by plasmatic concentrations. | 9 years
appearance auto-antibody and correlate to the clinical data | 9 years

CONTACTS AND LOCATIONS:
Overall Officials: Henri ROCHE, Pr, Principal Investigator — Institut Claudius Regaud
Locations (24):
- France (24):
  - Clinique Calabet, Agen
  - Clinique Claude Bernard, Albi
  - Centre Hospitalier d'Auch, Auch
  - CHU de Bordeaux, Bordeaux
  - Clinique Tivoli, Bordeaux
  - Institut Bergonié, Bordeaux
  - Polyclinique Bordeaux Nord, Bordeaux
  - Centre Hospitalier de Brive, Brive-la-Gaillarde
  - Centre Hospitalier de Cahors, Cahors
  - Centre Hospitalier Intercommunal de Castres-Mazamet, Castres
  - Hôpital Dupuytren CHU Limoges, Limoges
  - Centre Hospitalier de Mont de Marsan, Mont-de-Marsan
  - Centre Hospitalier de Montauban, Montauban
  - Centre Val d'Aurelle, Montpellier
  - Hôpital Caremeau CHU Nîmes, Nîmes
  - Centre Hospitalier de Pau, Pau
  - Centre Catalan d'Oncologie, Perpignan
  - Centre Hospitalier de Rodez, Rodez
  - Polyclinique de l'Ormeau, Tarbes
  - Claudius Regaud, Toulouse
  - CHU de Rangueil, Toulouse
  - Clinique Pasteur - Département d'Oncologie Médicale, Toulouse
  - Clinique Pasteur - Département de Radiothérapie, Toulouse
  - Clinique Saint-Jean du Languedoc, Toulouse

REFERENCES:
- [Derived] Puszkiel A, Dalenc F, Tafzi N, Marquet P, Debled M, Jacot W, Venat-Bouvet L, Ferrer C, Levasseur N, Paulon R, Dauba J, Evrard A, Mauries V, Filleron T, Chatelut E, Thomas F, White-Koning M. Identification of non-adherence to adjuvant letrozole using a population pharmacokinetics approach in hormone receptor-positive breast cancer patients. Eur J Pharm Sci. 2024 Aug 1;199:106809. doi: 10.1016/j.ejps.2024.106809. Epub 2024 May 22. PMID 38788907
- [Derived] Puszkiel A, Arellano C, Vachoux C, Evrard A, Le Morvan V, Boyer JC, Robert J, Delmas C, Dalenc F, Debled M, Venat-Bouvet L, Jacot W, Dohollou N, Bernard-Marty C, Laharie-Mineur H, Filleron T, Roche H, Chatelut E, Thomas F, White-Koning M. Model-Based Quantification of Impact of Genetic Polymorphisms and Co-Medications on Pharmacokinetics of Tamoxifen and Six Metabolites in Breast Cancer. Clin Pharmacol Ther. 2021 May;109(5):1244-1255. doi: 10.1002/cpt.2077. Epub 2020 Nov 10. PMID 33047329